CLINICAL TRIAL: NCT05641740
Title: Clinical Effects of a Single-session of Radiofrequency on Vascular Response and Pain Thresholds in Patients With Fibromyalgia: a Randomized Clinical Trial
Brief Title: Clinical Effects of Radiofrequency in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Research and teaching staff of the University of Granada, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RADIO-Fibromyalgia
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
Keywords: Radiofrequency Therapy; Peripheral blow flow; Core body temperature; Pain; Central sensitization; Peripheral nervous system; Thermography
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency Therapy Group (Experimental): The experimental group will receive a single-session of radiofrequency in their hands that has vasodilator action.
  Interventions: Device: Single-session of Radiofrequency
- Placebo Comparator: Control Group (Placebo Comparator): The placebo group will receive a single placebo radiofrequency session with the machine in pause mode.
  Interventions: Device: Control Placebo single-session of Radiofrequency

INTERVENTIONS:
Device: Single-session of Radiofrequency — The experimental group continue with their usual conservative and pharmacological treatment and will receive a single-session of monopolar dielectric capacitive radiofrequency in their hands. An Biotronic Advance Develops® (ABD-S25v) with a carrier wave frequency of 800-900 KHz of 850 KHz will be used. Patients will be placed in a seated position, with the forearms supinated and resting on a wooden table. An almond oil conductor will be applied to the hands. The application will be carried out with a circular head of 5 cm2 and for a total of 10 minutes on each of the palms of the hands.
  They will be evaluated at baseline and post-session.
  Other Names: Electric Stimulation Therapy
  Arms: Radiofrequency Therapy Group
Device: Control Placebo single-session of Radiofrequency — The control placebo group continue with their usual conservative and pharmacological treatment and will receive a placebo single-session of radiofrequency. This group will follow the same protocol and treatment time, but they will receive a placebo treatment (the device remains in paused mode), so that radiofrequency will not be applied.
  They will be evaluated at baseline and post-session.
  Other Names: Control Placebo Group
  Arms: Placebo Comparator: Control Group

SUMMARY:
The aim of this study is to analyze the effects of a single-session of Radiofrequency in patients with Fibromyalgia in comparison to a placebo group.

DETAILED DESCRIPTION:
The aim of this study is to analyze the effects of a single-session of Radiofrequency on peripheral vascular blood flow of the skin of the hands and core body temperature in patients with Fibromyalgia in comparison to a placebo group. Also, to study the clinical effects of the intervention on subjective pain perception, pain threshold to pressure and electrical pain threshold and intensity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia in accordance with the American College of Rheumatology criteria for classifying Fibromyalgia (2016 revision) by a rheumatologist of the Public Health System of Andalusia (Spain)
* Age from 18 to 70 years
* No other rheumatic diseases
* Absence of regular physical activity
* Limitation of usual activities due to pain on at least 1 day out of the previous 30

Exclusion Criteria:

* Male sex
* Presence of cardiac, renal or hepatic insufficiency;
* Severe physical disability
* Pregnancy or lactation
* Active infections
* Psychiatric illness
* Active tumor.
* Treatment with vasoactive drugs or anticoagulants or a history of drug use
* Skin disorders
* Any other non-pharmacological therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Peripheral vascular blood flow | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline temperature in the infrared thermography of the hands as indirect measure of peripheral vascular blood flow

SECONDARY OUTCOMES:
Pain Intensity: Visual Analog Scale | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline in pain in the Visual Analog Scale. Score range between 0-10 cm where 0 is in considered no pain and 10 is the worst pain imaginable.
Pain Threshold Electric Score | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline in the pain threshold electric score. We use the Pain Matcher a device that applied an electric current among the thumb and index finger with three recordings for pain threshold with a score ranging from 0 to 60
Pain Intensity Electric Score | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline in the pain intensity electric score. We use the Pain Matcher a device that applied an electric current among the thumb and index finger with three recordings for pain intensity with a score ranging from 0 to 60
Pressure Pain Threshold | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline un pressure pain threshold. A digital pressure algometer will be use to measure the pressure pain threshold bilaterally over 11 tender points considered by the American College of Rheumatology for Fibromyalgia diagnosis
Core body temperature | At the end of the radiofrequency session, an average of 20 minutes
  Change from baseline in core body temperature in patients with Fibromyalgia

CONTACTS AND LOCATIONS:
Overall Officials: Mª Encarnación ME Aguilar Ferrándiz, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Andalusia, Spain